CLINICAL TRIAL: NCT05167058
Title: Confirmatory Clinical Investigation of Electrocardiographic Diagnostic Performance of the Apple Watch Augmented With an Artificial Intelligence Algorithm
Brief Title: Electrocardiographic Diagnostic Performance of the Apple Watch Augmented With an Artificial Intelligence Algorithm
Status: Completed | Type: Observational
Sponsor: Cardiologs Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: SWAF
Record Dates: First submitted 2021-12-08; First posted 2021-12-22 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation; Tachycardia; Bradycardia; Premature Supraventricular Beat; Premature Ventricular Contraction
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia; Bradycardia; Atrial Premature Complexes; Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Cardiologs Platform — Smartwatch recordings interpreted by Cardiologs AI done simultaneously with each 12-lead ECG
  Other Names: Smartwatch

SUMMARY:
The SWAF study will compare the performance of a smartwatch combined with Cardiologs Platform algorithm in the detection of Atrial Fibrillation and other arrhythmias with that measured on a manually read 12-lead ECG in subjects hospitalized for cardioversion or AF ablation.

DETAILED DESCRIPTION:
The SWAF study is a prospective, non-significant risk, non-randomized, multicentric, open, comparative, confirmatory study.

Under subject consent, subjects hospitalized for cardioversion or AF ablation will have a smartwatch ECG recording done simultaneously with 12-lead ECG measurement right before the intervention. If a subject is found in Normal Sinus Rhythm he/she will be discharged otherwise the patient will undergo cardioversion and will have simultaneous recordings done a second time after the intervention. All the measurements will be done in accordance with the existing subject monitoring protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18, able and willing to participate in the study
* Subjects who are admitted to the hospital for a cardioversion or AF ablation procedure.
* Subjects having read the patient information letter and provided his/her consent to participate in writing, by dating and signing the informed consent prior to any trial-related procedure being conducted

Exclusion Criteria:

* Subjects with paced rhythm or implanted electronic devices
* Pregnant or breast-feeding subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 subjects: subjects who are hospitalized for cardioversion or AF ablation procedure per standard of care
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the performance of smartwatch ECG interpreted by Cardiologs Artificial Intelligence in detecting AF (Atrial Fibrillation or Flutter) as identified by the physician on the 12-lead ECG | Readings taken simultaneously right before and right after the cardioversion according to the monitoring protocol at the hospital
  Evaluation of the performance of smartwatch ECG interpreted by Cardiologs Artificial Intelligence in detecting AF (Atrial Fibrillation or Flutter) as identified by the physician on the 12-lead ECG in the independent annotation center, providing the ground truth from the 12-lead ECG

SECONDARY OUTCOMES:
Evaluation of the performance of smartwatch ECG interpreted by Cardiologs Artificial Intelligence in detecting AF as identified by the physician on the smartwatch ECG | Readings taken simultaneously right before and right after the cardioversion according to the monitoring protocol at the hospital
  Evaluation of the performance of smartwatch ECG interpreted by Cardiologs Artificial Intelligence in detecting AF as identified by the physician on the smartwatch ECG in the independent annotation center, providing the ground truth from the smartwatch ECG.
Evaluation of the performance of smartwatch ECG interpreted by Cardiologs Artificial Intelligence in detecting Sinus Rhythm as identified by the physician on the smartwatch ECG | Readings taken simultaneously right before and right after the cardioversion according to the monitoring protocol at the hospital
  Evaluation of the performance of smartwatch ECG interpreted by Cardiologs Artificial Intelligence in detecting Sinus Rhythm as identified by the physician on the smartwatch ECG in the independent annotation center, providing the ground truth from the smartwatch ECG.
Evaluation of the performance of smartwatch ECG interpreted by Cardiologs Artificial Intelligence in detecting Tachycardia as identified by the physician on the smartwatch ECG | Readings taken simultaneously right before and right after the cardioversion according to the monitoring protocol at the hospital
  Evaluation of the performance of smartwatch ECG interpreted by Cardiologs Artificial Intelligence in detecting Tachycardia as identified by the physician on the smartwatch ECG in the independent annotation center, providing the ground truth from the smartwatch ECG.
Evaluation of the performance of smartwatch ECG interpreted by Cardiologs Artificial Intelligence in detecting Bradycardia as identified by the physician on the smartwatch ECG | Readings taken simultaneously right before and right after the cardioversion according to the monitoring protocol at the hospital
  Evaluation of the performance of smartwatch ECG interpreted by Cardiologs Artificial Intelligence in detecting Bradycardia as identified by the physician on the smartwatch ECG in the independent annotation center, providing the ground truth from the smartwatch ECG.
Evaluation of the performance of smartwatch ECG interpreted by Cardiologs Artificial Intelligence in detecting Premature Supraventricular Complexes as identified by the physician on the smartwatch ECG | Readings taken simultaneously right before and right after the cardioversion according to the monitoring protocol at the hospital
  Evaluation of the performance of smartwatch ECG interpreted by Cardiologs Artificial Intelligence in detecting Premature Supraventricular Complexes as identified by the physician on the smartwatch ECG in the independent annotation center, providing the ground truth from the smartwatch ECG.
Evaluation of the performance of smartwatch ECG interpreted by Cardiologs Artificial Intelligence in detecting Premature Ventricular Complexes as identified by the physician on the smartwatch ECG | Readings taken simultaneously right before and right after the cardioversion according to the monitoring protocol at the hospital
  Evaluation of the performance of smartwatch ECG interpreted by Cardiologs Artificial Intelligence in detecting Premature Ventricular Complexes as identified by the physician on the smartwatch ECG in the independent annotation center, providing the ground truth from the smartwatch ECG.
Assessment of the proportion of smartwatch ECGs identified as inconclusive by Cardiologs Artificial Intelligence and by the physician | Readings taken simultaneously right before and right after the cardioversion according to the monitoring protocol at the hospital
  Assessment of the proportion of smartwatch ECGs identified as inconclusive by Cardiologs Artificial Intelligence and by the physician. Inconclusive may mean that there may have been too much artefact or noise to acquire a good signal or that the rhythm is unclassifiable or contains other abnormal rhythm.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Y Wan, MD, Principal Investigator — Columbia University, New York
Locations (3):
- United States (3):
  - Hackensack Meridian School of Medicine, Hackensack, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Columbia University Medical Center/ NewYork Presbyterian Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No